CLINICAL TRIAL: NCT01357629
Title: Observational Follow-up Extension Study to Evaluate Long-term Safety and Tolerability of Immunizations With AFFITOPE AD02 Applied During AFFiRiS002 and AFF004A in Patients With Alzheimer's Disease
Brief Title: Observational Follow-up Extension Study of AFF002 and AFF004A in Patients With Alzheimer's Disease
Status: Terminated | Type: Observational
Why Stopped: The Study could not be done for every potential participant as planned in the protocol for organizational reasons.
Sponsor: Affiris AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AFF004E
Record Dates: First submitted 2011-03-21; First posted 2011-05-23 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Alzheimer´s Disease
Keywords: Vaccination follow-up

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
This study examines the long term Safety Follow-up of first patients vaccinated with AD02.

DETAILED DESCRIPTION:
Patients who have received AD02 during AFF002 and AFF004A will be observed.

ELIGIBILITY:
Inclusion Criteria:

* participation in AFF002 and AFF004A

Exclusion Criteria:

* no vaccination with AD02

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Alzheimer´s Disease
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2011-07; Primary Completion 2013-04 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety | up to 2 years
  collection and evaluation of AEs, SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Achim Schneeberger, MD, Study Director — Sponsor GmbH; Siegfried Kasper, MD, Principal Investigator — Medical University Vienna
Locations (2):
- Austria (2):
  - Studienzentrum der PROSENEX Ambulatoriumsbetriebs GmbH, Vienna, Vienna
  - Univ. Klinik für Psychiatire und Psychotherapie, Vienna